CLINICAL TRIAL: NCT02880189
Title: Combined Endoscopic Ultrasound Guided Core Liver Biopsy and Intragastric Balloon Placement for the Diagnosis and Management of Nonalcoholic Steatohepatitis and Obesity
Brief Title: EUS Guided Core Liver Biopsy and IGB Placement for the Diagnosis and Management of NASH and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barham K. Abu Dayyeh, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-009262
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Obesity; Non-Alcoholic Steatohepatitis
Keywords: Non-Alcoholic Steatohepatitis (NASH); NASH with Fibrosis; Intragastric Balloon; Orbera; Orbera Intragastric Balloon
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Other): All subjects will be receiving the Orbera Intragastric Balloon and will be undergoing Endoscopic Ultrasound guided core liver biopsy.
  Interventions: Device: Orbera Intragastric Balloon; Procedure: Endoscopic Ultrasound Guided Core Liver Biopsy

INTERVENTIONS:
Device: Orbera Intragastric Balloon — The Orbera Intragastric Balloon will be placed in the stomach endoscopically through a catheter under conscious sedation. The procedure takes about 20 minutes to complete. The balloon will stay in place for 6 months and then it will be removed endoscopically.
Procedure: Endoscopic Ultrasound Guided Core Liver Biopsy

SUMMARY:
This study is designed to investigate the impact of weight loss achieved with the IGB on NASH with early fibrosis in a select cohort of patients with obesity preselected to have a high pre-test probability of having NASH with early fibrosis based on magnetic resonance elastography (MRE)-Hepatogram. In addition, this study will explore potential non-invasive imaging criteria for NASH and early fibrosis using EUS-Elastography.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Non-alcoholic Steatohepatitis with early evidence of fibrosis as seen on MRE-hepatogram
* Referred clinically for an intragastric balloon placement for weight loss

Exclusion Criteria:

* Women who are pregnant or plan to be pregnant or are breastfeeding
* Previous history of gastric surgery
* Current or recent (within 6 months) gastric or duodenal ulcers
* Gastroparesis
* Liver cirrhosis
* Coagulopathy or active use of coagulation
* Inability to provide a written informed consent

Ages: 22 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barham Abu Dayyeh, M.D., Principal Investigator — Mayo Clinic

REFERENCES:
- [Derived] Bazerbachi F, Vargas EJ, Rizk M, Maselli DB, Mounajjed T, Venkatesh SK, Watt KD, Port JD, Basu R, Acosta A, Hanouneh I, Gara N, Shah M, Mundi M, Clark M, Grothe K, Storm AC, Levy MJ, Abu Dayyeh BK. Intragastric Balloon Placement Induces Significant Metabolic and Histologic Improvement in Patients With Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2021 Jan;19(1):146-154.e4. doi: 10.1016/j.cgh.2020.04.068. Epub 2020 Apr 30. PMID 32360804
- [Derived] Bazerbachi F, Vargas EJ, Matar R, Storm AC, Mounajjed TM, Topazian MD, Levy MJ, Chandrasekhara V, Abu Dayyeh BK. EUS-guided core liver biopsy sampling using a 22-gauge fork-tip needle: a prospective blinded trial for histologic and lipidomic evaluation in nonalcoholic fatty liver disease. Gastrointest Endosc. 2019 Dec;90(6):926-932. doi: 10.1016/j.gie.2019.08.006. Epub 2019 Aug 19. PMID 31437454
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Single: All subjects will be receiving the Orbera Intragastric Balloon and will be undergoing Endoscopic Ultrasound guided core liver biopsy.
  Orbera Intragastric Balloon: The Orbera Intragastric Balloon will be placed in the stomach endoscopically through a catheter under conscious sedation. The procedure takes about 20 minutes to complete. The balloon will stay in place for 6 months and then it will be removed endoscopically.
  Endoscopic Ultrasound Guided Core Liver Biopsy
Period: Overall Study
Arm/Group | Single
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 54 [34 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21
Body Mass Index [Median (Full Range); unit: kg/m^2] | 44 [32 to 55]

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss Achieved With Intragastric Balloon (IGB)
Description: Total number of subjects with two points or greater improvement on objective Non-alcoholic Steatohepatitis (NASH) histopathological parameters. The NAS scale can range from 0 to 8 and is calculated by the sum of scores of steatosis (0-3), lobular inflammation (0-3) and hepatocyte ballooning (0-2).
Time Frame: Baseline to 6 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 21
Participants | 17

2. Secondary Outcome: Diagnosis of NASH and Early Fibrosis by Endoscopic Ultrasound (EUS) Guided Liver Core Biopsies
Description: Total number of subjects correctly diagnosed with NASH and Early Fibrosis by EUS guided core liver biopsies
Time Frame: Baseline to 6 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 21
Participants | 21

ADVERSE EVENTS:
Time Frame: The study treatment follow-up period was defined from enrollment in the study to 6 months after balloon removal.
Arm/Group | Single
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=21)
Epigastric pain (Gastrointestinal disorders) | 3 (3)
Laryngospasm (General disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Non-ST-elevation myocardial infarction (NSTEMI) (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT02880189/Prot_SAP_000.pdf